CLINICAL TRIAL: NCT02569788
Title: Phase I/II Trail Evaluating Carbon Ion Radiotherapy for Salvaging Treatment of Locally Recurrent Nasopharyngeal Carcinoma
Brief Title: Trail Evaluating Carbon Ion Radiotherapy for Locally Recurrent Nasopharyngeal Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual of patients.
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Jiade J. Lu, Professor, Shanghai Proton and Heavy Ion Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-HNCNS-2015-01
Record Dates: First submitted 2015-10-01; First posted 2015-10-07 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: re-irradiation; carbon ion radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Heavy Ion Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CIRT Arm (Experimental): Patients included in this arm were treated with carbon ion radiotherapy (CIRT).
  Interventions: Radiation: Carbon ion radiotherapy (CIRT)

INTERVENTIONS:
Radiation: Carbon ion radiotherapy (CIRT) — Five dose levels (55GyE, 57.5GyE, 60GyE, 62.5GyE, 65GyE) are planned within the Phase I part. Daily fraction of 2.5 GyE will be delivered for all dose levels. After the recommended dose (RD), i.e., MTD, is determined or if the treatments to 65 GyE are safely delivered, the recommended dose (or 65 GyE) will be the prescribed dose in the Phase II part of the study. Ninty-five percent (95%) of the isodose line should cover the GTV+3~5mm.

SUMMARY:
The purpose of this study is to determine the maximal tolerated dose (MTD) of re-irradiation using carbon ion radiotherapy (CIRT) in the treatment of locally recurrent nasopharyngeal cancer (NPC) and to evaluate the efficacy of such treatment at the MTD. Participants will be treated with CIRT with escalating dose regimens to evaluate the maximal tolerated dose (MTD) in terms of acute and subactue toxicity observed during and within 4 months after the completion of CIRT. Once the MTD for locally recurrent NPC is determined, the MTD will be used as the recommended dose to patients fulfilling the inclusion criteria in the Phase II part of the trial.

DETAILED DESCRIPTION:
The purpose of this study is to determine the maximal tolerated dose (MTD) of re-irradiation using carbon ion radiotherapy (CIRT) in the treatment of locally recurrent nasopharyngeal cancer (NPC) and to evaluate the efficacy of such treatment at the MTD. Participants will be treated with CIRT with escalating dose starting from 55GyE (2.5GyE/daily fraction) to potentially 65GyE (2.5GyE/daily fraction) to evaluate the maximal tolerated dose (MTD) in terms of acute and subactue toxicity observed during and within 4 months after the completion of CIRT. Time-to-event continual reassessment method (TITE-CRM) is used for the phase I dose escalating part of the trial and approximately 25 patients will be accrued. Once the MTD for locally recurrent NPC is determined, the MTD will be used as the recommended dose to patients fulfilling the inclusion criteria in the Phase II part of the trial. The Phase II part of the trial will be a single phase single arm study.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed NPC
* Completed a definitive course of intensity-modulated photon radiation therapy (IMXT) to a total dose of ≥ 66 Gy
* Recurrence diagnosed more than 12 months after the initial course of IMXT
* Age ≥ 14 and < 70 years of age
* Karnofsky Performance Score ≥70
* Willing to accept adequate contraception for women with childbearing potential
* Ability to understand character and individual consequences of the clinical trial
* Willing to sign the written informed consent; Informed consent must be signed before the enrollment in the trial

Exclusion Criteria:

* Local recurrence of NPC diagnosed within 12 months from the completion of previous course of radiation therapy
* Presence of distant metastasis
* Technology used other than IMXT (including brachytherapy following IMXT) for the treatment of initial diagnosis of NPC
* Pregnant or lactating women
* Patients who have not yet recovered from acute toxicities of prior therapies
* A diagnosis of malignancy other than CIS of the cervix, BCC and SCC of the skin within the past 5 years
* Refusal of the patient to participate into the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Time interval from the start of CIRT to 4 months after the completion of CIRT

SECONDARY OUTCOMES:
Overall survival of all patients | From the diagnosis of local recurrence of NPC, a median of 2 years
Progression-free survival of all patients | From the completion of CIRT, a median of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jiade J Lu, MD, Principal Investigator — Shanghai Proton and Heavy Ion Center,Shanghai, SPHIC
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, Shanghai Municipality, China